CLINICAL TRIAL: NCT02826356
Title: Efficient Treatments for ACE-I and ARB-induced Angioedema Exist and Should be Available to All Patients. Analysis of Their Availability and Influencing Factors in the Area Around Lyon, France
Brief Title: Analysis of the Availability of the Treatments for ACE-I and ARB-induced Angioedema
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0430
Record Dates: First submitted 2016-07-05; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: ACE-I and ARB-induced Angioedema.
Keywords: Angioedema; Emergency treatment; Treatment availability; Health Equity
MeSH Terms: conditions — Angioedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Specific treatments for angiotensin-converting-enzyme inhibitor (ACE-I) and angiotensin-receptor-blocker (ARB)-induced angioedema exist. Early access to these treatments is challenging because they are expensive and have short shelf lives making it illusory that all emergency department (ED) stock them. The aim of this retrospective study was to define, for each patient with a confirmed ACE-I or ARB-induced angioedema, at which step of the care, the specific treatment was administered. The second objective was to analyse the availability of these treatment in the area around Lyon, France and the factors that may influence it.

ELIGIBILITY:
Inclusion Criteria:

* Every patient followed for the first time in our reference center for severe confirmed ACE-I or ARB-induced angioedema. Data were analyzed from patients attended either in a specialized angioedema consultation or during a hospitalization in our intensive care unit.
* Severe attack was defined either by its localization over the shoulder or by an severe abdominal attack.

Exclusion Criteria:

- Patients which received no specific treatment (icatibant, C1-inhibitor concentrate) were excluded.

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with a specific treatment for bradykinin-mediated angioedema for a severe attack of angioedema due to ACE-inhibitors or ARB during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2016-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Step of the care allowing the patients to benefit from a specific treatment. | October 2010 to December 2014
  Three answers are possible. Patients were treated with the specific medication (icatibant or C1-inhibitor concentrate) either in the first ED or by the medical ambulance team, or by the investigators reference center's intensive care unit.

SECONDARY OUTCOMES:
Epidemiological characteristics | October 2010 to December 2014
  The investigators collect data such as age, sex, localization of the angioedema.
Triggering treatments | October 2010 to December 2014
  The investigators detail which ACE-inhibitor, which ARB and eventually which co-medication was taken and triggered the angioedema.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard FLOCCARD, MD, Principal Investigator — Hospices Civils de Lyon, Département d'Anesthésie-Réanimation, Hôpital Edouard Herriot, Lyon, France.
Locations (1):
- Hospices Civils de Lyon, Département d'Anesthésie-Réanimation, Hôpital Edouard Herriot, Lyon, France., Lyon, France